CLINICAL TRIAL: NCT02986191
Title: Clinical Applications of 3D Collagen Matrix (Mucograft®) in the Management of Gingival Recession: a Randomized Controlled Trial
Brief Title: The Use of Mucograft® to Treat Gingival Recession
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Perio-01-2016
Record Dates: First submitted 2016-11-29; First posted 2016-12-08 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Gingival Recession
Keywords: gingival graft; free gingival graft; coronally advanced flap; reduced keratinized gingiva
MeSH Terms: conditions — Gingival Recession | interventions — Mucograft

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mucograft (Experimental): One side of the mouth will be subjected to Mucograft in this split-mouth study design.
  Interventions: Procedure: Mucograft
- Connective tissue graft (Active Comparator): The opposite side of the mouth will be subjected to a connective tissue graft.
  Interventions: Procedure: Connective Tissue Graft

INTERVENTIONS:
Procedure: Mucograft — This method of grafting will be used to treat the gingival recession using coronally advanced flaps.
  Arms: Mucograft
Procedure: Connective Tissue Graft — This will be used in the traditional manner to correct gingival recession
  Arms: Connective tissue graft

SUMMARY:
Twenty patients with gingival recession will be enrolled in this trial. Gingival recession will be treated in one side by applying Mucograft® with coronally advanced flap (CAF) while on the opposite side a connective tissue graft (from the palate) will be applied with a CAF.

Patients will be followed for 3 and 6 months by measuring the clinical indexes and statistical analyses will be performed to compare the results and to assess the success of Mucograft®.

DETAILED DESCRIPTION:
Many surgical techniques have used to treat gingival recession such aas repositioned flaps, autologous soft tissue grafts (connective tissue graft or free gingival grafts) or allografts like acellular dermal which can be used as substitutes for palatal donor tissue. Mucograft® (3D collagen matrix) is also an allograft from porcine origin and is designed for soft tissue regeneration and considered the ideal solution to autogenous soft tissue grafts and it provides an ideal matrix for blood vessel and soft tissue ingrowth.

ELIGIBILITY:
Inclusion Criteria:

* Presence of Type I or II (Miller Classification) of gingival recession

Exclusion Criteria:

* Smoking
* Pregnancy or lactating
* Presence of any systematic diseases can affect the periodontal surgery.
* Subjects with significant moderate to severe periodontal disease.
* Patients under orthodontic treatment
* Presence of restorative materials (e.g. crown)
* Effectiveness of frenum
* Subjects have failed to maintain good plaque control.
* Subjects having previous surgical treatment for covering the recession in the chosen area.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Change in the Clinical Attachment Level Index | Measurements will be done at :(1) one hour before applying the graft, (2) at three months exactly post-operatively and (3) at six months exactly post-operatively
  Clinical Attachment Level is dependent on measuring the pocket depth as well as the amount of gingival recession using specific tools. The measurement is going to be recorded in millimeters.

SECONDARY OUTCOMES:
Change in Probing Depth | Measurements will be done at :(1) one hour before applying the graft, (2) at three months exactly post-operatively and (3) at six months exactly post-operatively
  Probing depth is going to be measuring using a specific tool (UNC-15 probe).
Change in Gingival Recession | Measurements will be done at :(1) one hour before applying the graft, (2) at three months exactly post-operatively and (3) at six months exactly post-operatively
  Gingival recession is measured from the cemento-enamel junction to the gingival margin of the recessed tissues.
Change in Gingival Biotype | Measurements will be done at :(1) one hour before applying the graft, (2) at three months exactly post-operatively and (3) at six months exactly post-operatively
  Gingival biotype is assessed by an endodontic file which used to determine the thickness of the gingival tissues (i.e. thick or thin).
Change in Root Coverage Index | Measurements will be done at :(1) one hour before applying the graft, (2) at three months exactly post-operatively and (3) at six months exactly post-operatively
  The amount of root exposure will be measured and compared to the total length of the root
Change in Resistance to Muscular Pull | Measurements will be done at :(1) one hour before applying the graft, (2) at three months exactly post-operatively and (3) at six months exactly post-operatively
  The cheeks or lips are going to be retracted by hand or by a mirror in order to see the movement of the free gingival tissues. The movement will be esitmated in millimeters.
Change in Color Match Index | Measurements will be done at :(1) one hour before applying the graft, (2) at three months exactly post-operatively and (3) at six months exactly post-operatively
Shrinkage index at three months | Measurements will be done at two time points to calculate the amount of shrinkage :(1) at one hour before applying the graft, (2) at three months exactly post-operatively.
Shrinkage index at six months | Measurements will be done at two time points to calculate the amount of shrinkage :(1) at one hour before applying the graft, (2) at six months exactly post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Haydar Barakat, DDS MSc, Principal Investigator — PhD Student in Periodontics, University of Damascus Dental School, Damascus, Syria; Suleiman Dayoub, DDS MSc PhD, Study Director — Associate Professor of Periodontics, Department of Peridontics, Univ. of Damascus Dental School
Locations (1):
- Department of Periodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herford AS, Akin L, Cicciu M, Maiorana C, Boyne PJ. Use of a porcine collagen matrix as an alternative to autogenous tissue for grafting oral soft tissue defects. J Oral Maxillofac Surg. 2010 Jul;68(7):1463-70. doi: 10.1016/j.joms.2010.02.054. Epub 2010 Apr 22. PMID 20417009
- [Background] Nevins M, Nevins ML, Kim SW, Schupbach P, Kim DM. The use of mucograft collagen matrix to augment the zone of keratinized tissue around teeth: a pilot study. Int J Periodontics Restorative Dent. 2011 Jul-Aug;31(4):367-73. PMID 21837302
- [Background] Rocchietta I, Schupbach P, Ghezzi C, Maschera E, Simion M. Soft tissue integration of a porcine collagen membrane: an experimental study in pigs. Int J Periodontics Restorative Dent. 2012 Feb;32(1):e34-40. PMID 22254233
- [Background] Cardaropoli D, Tamagnone L, Roffredo A, Gaveglio L. Treatment of gingival recession defects using coronally advanced flap with a porcine collagen matrix compared to coronally advanced flap with connective tissue graft: a randomized controlled clinical trial. J Periodontol. 2012 Mar;83(3):321-8. doi: 10.1902/jop.2011.110215. Epub 2011 Jul 1. PMID 21721988
- [Background] Jepsen K, Jepsen S, Zucchelli G, Stefanini M, de Sanctis M, Baldini N, Greven B, Heinz B, Wennstrom J, Cassel B, Vignoletti F, Sanz M. Treatment of gingival recession defects with a coronally advanced flap and a xenogeneic collagen matrix: a multicenter randomized clinical trial. J Clin Periodontol. 2013 Jan;40(1):82-9. doi: 10.1111/jcpe.12019. Epub 2012 Oct 10. PMID 23050490
- [Background] McGuire MK, Scheyer ET. Randomized, controlled clinical trial to evaluate a xenogeneic collagen matrix as an alternative to free gingival grafting for oral soft tissue augmentation. J Periodontol. 2014 Oct;85(10):1333-41. doi: 10.1902/jop.2014.130692. Epub 2014 Mar 5. PMID 24597764
- [Background] McGuire MK, Scheyer ET. Long-Term Results Comparing Xenogeneic Collagen Matrix and Autogenous Connective Tissue Grafts With Coronally Advanced Flaps for Treatment of Dehiscence-Type Recession Defects. J Periodontol. 2016 Mar;87(3):221-7. doi: 10.1902/jop.2015.150386. Epub 2015 Oct 15. PMID 26469812